CLINICAL TRIAL: NCT00031031
Title: Phase I Study of KLT in Patients With Solid Tumors Refractory to Standard Therapy
Brief Title: Kanglaite Injection Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KangLaiTe USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN-001-01
Record Dates: First submitted 2002-02-20; First posted 2002-02-22 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Solid Tumors Refractory To Standard Therapy; Neoplasms
Keywords: MTD; Safety; Pharmacokinetics; Efficacy
MeSH Terms: conditions — Neoplasms | interventions — kang-lai-te

INTERVENTIONS:
Drug: Kanglaite Injection (KLT)

SUMMARY:
The Kanglaite Injection (KLT)is a novel broad spectrum anti-cancer injection produced from traditional Chinese medicinal herbs (the Coix Seed). It was approved in China in 1995 and has become the most popular anti-cancer drug in China. In June of 2001, the Phase I study of KLT commenced at the Huntsman Cancer Institute in Salt Lake City, Utah, with the objectives of 1) To determine the maximum tolerated dose (MTD) and the safety profile of KLT in patients with refractory solid tumors; 2) To determine the pharmacokinetics of KLT in patients with refractory solid tumors; and 3) To gather preliminary efficacy data. The method of testing is open-label, sequential cohort, dose-escalation study.

ELIGIBILITY:
* Patients with histological evidence of malignancy that has become refractory to standard therapy, or for whom effective standard therapy does not exist.
* Patients with an estimated life-expectancy of at least 3 months
* Patients with a Karnofsky Performance Score of at least 60%
* Patients with no history of congestive heart failure (CHF), and normal ejection fraction by echocardiography
* Patients with adequate renal and hepatic function
* Patients with adequate bone marrow status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2001-06; Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Wheeler, M.D., Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institue, Salt Lake City, Utah, United States